CLINICAL TRIAL: NCT07016828
Title: Comparing Accuracy of Pterygoid Implants Placement Using Computer-guided Surgical Templates Versus Free Hand Technique
Brief Title: Guided Pterygoid Implant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Norhan Magdy Ahmed Yousef, dentist in medical administration at fayoum university, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pterygoid implant
Record Dates: First submitted 2025-06-03; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Atrophy of the Posterior Maxilla
Keywords: guided surgery; pterygoid implant; atrophic maxilla
MeSH Terms: conditions — Atrophic Maxilla

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Surgery group (Active Comparator): Implants placed using CBCT-based 3D surgical guides.
  Interventions: Device: guided surgery technique
- free hand technique group (Placebo Comparator): Freehand placement based on anatomical landmarks.
  Interventions: Procedure: Free hand technique

INTERVENTIONS:
Device: guided surgery technique — * Clinical examination will be performed and preoperative CBCT will be taken for all the patients prior to the surgery to evaluate the posterior maxilla for the placement of the pterygoid implants.
  * Ideal pterygoid implant placement will be planned using the BlueSky Bio software (USA) which will be mostly to emerge from the third molar position and to engage the dense pillar of bone formed by the pyramidal process and pterygoid process of sphenoid bone.
  * surgical guide will be fabricated which will be either soft tissue without flap elevation.
  Arms: Guided Surgery group
Procedure: Free hand technique — the surgery will be done without the use of the surgical guides depending on the anatomical landmarks.
  Arms: free hand technique group

SUMMARY:
Introduction & Background Alveolar ridge resorption after tooth extraction leads to significant bone loss, complicating prosthetic rehabilitation. Traditional bone grafting methods, though effective, involve long healing times and risks. Pterygoid implants offer a graft-free alternative by engaging dense bone structures like the pterygoid process. However, their placement is technically challenging due to limited visibility and proximity to critical structures. Computer-guided surgery may improve accuracy and reduce complications compared to freehand techniques.

Research Question Does computer-guided surgery enhance the accuracy of pterygoid implant placement in atrophic maxillae compared to freehand techniques? Aim To compare the accuracy of computer-generated 3D surgical guides versus freehand placement of pterygoid implants.

Hypothesis

* H0: No difference in accuracy between techniques.
* Hₐ: there is difference between two techniques Study Design A prospective randomized controlled trial (1:1 allocation) with 12 implants (6 per group(.

Patient Selection Inclusion Criteria: Severe posterior maxillary atrophy (Cawood & Howell V-VI), residual bone height <4mm, age 21-75.

Exclusion Criteria: Contraindications for surgery, uncontrolled systemic diseases, or acute sinus infections.

Methods

* Group A: Implants placed using CBCT-based 3D surgical guides.
* Group B: Freehand placement based on anatomical landmarks.
* Primary Outcome: Implant position accuracy (postoperative CBCT vs. virtual plan(.
* Secondary Outcomes: Surgical time, complications, and stability. Surgical Procedure
* Osteotomy: Angled drilling (45-60°) into the pterygoid process.
* Implant Placement: Torque ≥30 Ncm for primary stability.
* Postoperative Care: Antibiotics, analgesics, and follow-up CBCT at one week. Statistical Analysis Data analyzed using SPSS, with G*Power determining sample size (85% power, α = 0.05(.

Ethical Considerations Approved by institutional review boards, with informed consent and confidentiality maintained.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severe posterior maxillary atrophy (Class V-VI Cawood & Howell classification) requiring pterygoid implant placement.
2. Patients with severe alveolar bone atrophy in posterior maxilla (Residual alveolar bone height <4mm in posterior maxilla precluding conventional implant placement).
3. Adequate interarch space ≥7mm for prosthetic rehabilitation.
4. Presence of pneumatized maxillary sinus with insufficient bone for sinus augmentation.
5. Patients aged 21-75 years with completed craniofacial growth.

Exclusion Criteria:

1. Patients with systemic conditions contra-indicating general anesthesia.
2. Patients with conditions contraindicating implant placement (e.g.:

   radiation to the head and neck, intra-venous bisphosphonates, uncontrolled Diabetes mellitus).
3. Patients with acute maxillary sinus infection or maxillary sinus cyst.
4. Restricted mouth opening (less than 3cm inter-arch distance anteriorly).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-07-30 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy of implant position | the patient will make postoperative CBCT after one week of the surgery to compare it with the preoperative virtual planning done on the preoperative CBCT.
  The primary outcome will be measured by comparing the position of implant in the virtual plan with that in the postoperative implant or the actual implant and this will be done by making a superimposition of the virtual plan with the postoperative CBCT then putting points on the coronal and apical parts of implants and then start to measure the following data:
  1. direct linear measurements between the coronal and apical points of the virtual and actual implants (measured in millimeters)
  2. angular deviations between the long axis of virtual and postoperative or actual implants.(measured in degrees)
  3. indirect measurements of the coronal and apical points of virtual and actual implants to 3d planes.(measured in mm)
  All of this will be done for both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
I still have no decision until i start my research and getting approvals from the patients to protect their right.